CLINICAL TRIAL: NCT01531283
Title: Impact of Unacylated Ghrelin on Beta-cell Function in Humans
Brief Title: Deacylated Ghrelin and Beta Cell Function
Acronym: UAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: David Dalessio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David Dalessio, Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 10-07-19-04; 1R03DK089090-01 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: the Diabetic Process
Keywords: unacylated ghrelin; beta cell function
MeSH Terms: interventions — acyl-ghrelin; ghrelin, des-n-octanoyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- decaylated ghrelin (Experimental): UAG (4.0 µg/kg/hr)
  Interventions: Drug: unacylated ghrelin
- acyl ghrelin (Experimental): AG (1.0 µg/kg/hr)
  Interventions: Drug: acyl ghrelin
- combined acyl and desacyl ghrelin (Experimental): the combination of AG (1 µg/kg/hr) and UAG (4 µg/kg/hr)
  Interventions: Drug: combined acyl and desacyl ghrelin
- saline (Placebo Comparator): saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: unacylated ghrelin — IV, UAG (4.0 µg/kg/hr), one time, duration of study visit (approximately 5 hours)
  Arms: decaylated ghrelin
Drug: acyl ghrelin — IV, AG (1.0 µg/kg/hr), one time, duration of study visit (approximately 5 hours)
  Arms: acyl ghrelin
Drug: combined acyl and desacyl ghrelin — IV, the combination of AG (1 µg/kg/hr) and UAG (4 µg/kg/hr), one time, for the duration of the study visit (approximately 5 hours)
  Arms: combined acyl and desacyl ghrelin
Drug: saline — IV, saline, one time, for the duration of the study visit(approximately 5 hours)
  Arms: saline

SUMMARY:
Use of human unacylated ghrelin (UAG, also called des-octanoyl ghrelin) to study physiology in healthy subjects. The proposed research is an investigator-initiated study funded by the National Institutes of Health designed to examine the effect of physiologic levels of UAG on the regulation of glucose homeostasis as well as beta cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy men and women. Only premenopausal women who are using an adequate method of contraception at Screening and who agree to continue the contraception during the study will be included. Male subjects do not need to use on birth control.
2. Ages between 18 and 50 years, inclusive.
3. BMI between 18.5 and 29.9 kg/m2, inclusive

Exclusion Criteria:

1. History or clinical evidence of impaired fasting glucose or impaired glucose tolerance or diabetes mellitus, myocardial infarction, history or symptoms of congestive heart failure, history of cancer or anorexia nervosa, history or active liver or renal disease (AST or ALT >2x upper limits of normal, calculated glomerular filtration rate [GFR] <60).
2. A baseline resting systolic blood pressure of less than 100 mm Hg.
3. History of growth hormone deficiency or excess disorders (acromegaly, pituitary gigantism, panhypopituitarism); history of adrenal insufficiency or Cushing's disease/syndrome; history of neuroendocrine tumors.
4. Anemia defined as hematocrit <33%.
5. Use of medications that alter insulin sensitivity: niacin, glucocorticoids, metformin, thiazolidinediones, exenatide, or atypical anti-psychotics.
6. Pregnancy or lactation.
7. BMI <18 kg/m2 or BMI >30 kg/m2; fasting plasma glucose >100 mg/dl and/or 2 hr plasma glucose >140 mg/dl on a 75 g oral glucose tolerance test.
8. Electrocardiogram (ECG) abnormalities: specifically, myocardial ischemia, previous myocardial ischemia, atrial fibrillation, second or third degree heart block and complete right or left bundle branch block.
9. Females who are on progesterone-only contraception and those who have irregular menses.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
acute insulin release (AIRg) | one year
  The primary outcome measure will be AIRg. This is calculated as the incremental insulin release,following IV glucose administration. (For the first ten minutes of the study visit.)

SECONDARY OUTCOMES:
Insulin sensitivity | one year
  1. Insulin sensitivity is quantified as the insulin sensitivity index (SI) using Bergman's minimal model of glucose kinetics from the glucose and insulin results obtained from a FSIGT.
Disposition index | one year
  2. The disposition index (DI) is a measure of β-cell function. It accounts for the modulating effect of insulin sensitivity on β-cell responses. It is calculated as the product of the SI and AIRg
glucose tolerance | one year
  3. Glucose tolerance is measured by glucose disappearance constant. This is calculated as the slope of the natural log of glucose during the study visit, during a set time frame.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States